CLINICAL TRIAL: NCT04845633
Title: Evaluation of the Effectiveness of Customized Handle Toothbrush in Dental Plaque Control in Healthy Children and Children With Down Syndrome
Brief Title: Effectiveness of Customized Handle Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UDDS-Pedo-01-2021
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-06

CONDITIONS: Dental Plaque; Dental Prophylaxis; Dental Care
Keywords: Customized Handle Toothbrush; Dental Primary Prevention; Down Syndrome
MeSH Terms: conditions — Dental Plaque; Down Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy children using conventional toothbrush (Other)
  Interventions: Other: Evaluation of the Effectiveness of Conventional Toothbrush in Dental Plaque Control in Healthy Children
- Healthy children using toothbrush with Customized Handle (Experimental)
  Interventions: Other: Evaluation of the Effectiveness of Customized Handle Toothbrush in Dental Plaque Control in Healthy Children
- Children with Down syndrome using conventional toothbrush (Other)
  Interventions: Other: Evaluation of the Effectiveness of Conventional Toothbrush in Dental Plaque Control in Children with Down Syndrome
- Children with Down syndrome using toothbrush with Customized Handle (Experimental)
  Interventions: Other: Evaluation of the Effectiveness of Customized Handle Toothbrush in Dental Plaque Control in Children with Down Syndrome

INTERVENTIONS:
Other: Evaluation of the Effectiveness of Conventional Toothbrush in Dental Plaque Control in Healthy Children — Healthy children will be given conventional toothbrush.Plaque scores in groups will be assess pre-brushing and post-brushing in baseline, a week, and after 3 weeks by using the Turesky Modification of the Quigley-Hein Plaque Index (TMQHPI) for both buccal and lingual surfaces
  Arms: Healthy children using conventional toothbrush
Other: Evaluation of the Effectiveness of Customized Handle Toothbrush in Dental Plaque Control in Healthy Children — Healthy children will be given toothbrush with Customized Handle.Plaque scores in groups will be assess pre-brushing and post-brushing in baseline, a week, and after 3 weeks by using the Turesky Modification of the Quigley-Hein Plaque Index (TMQHPI) for both buccal and lingual surfaces
  Arms: Healthy children using toothbrush with Customized Handle
Other: Evaluation of the Effectiveness of Conventional Toothbrush in Dental Plaque Control in Children with Down Syndrome — Children with Down syndrome will be given conventional toothbrush.Plaque scores in groups will be assess pre-brushing and post-brushing in baseline, a week, and after 3 week by using the Turesky Modification of the Quigley-Hein Plaque Index (TMQHPI) for both buccal and lingual surfaces
  Arms: Children with Down syndrome using conventional toothbrush
Other: Evaluation of the Effectiveness of Customized Handle Toothbrush in Dental Plaque Control in Children with Down Syndrome — Children with Down syndrome will be given toothbrush with Customized Handle.Plaque scores in groups will be assess pre-brushing and post-brushing in baseline, a week, and after 3 weeks by using the Turesky Modification of the Quigley-Hein Plaque Index (TMQHPI) for both buccal and lingual surfaces
  Arms: Children with Down syndrome using toothbrush with Customized Handle

SUMMARY:
People with special needs suffer from many difficulties, including mental, physical or motor, which increase the difficulty of obtaining good oral health.

Therefore, some adjustments must be made to help these patients maintain oral health.

The aim of the current research is to modify the traditional toothbrush grip by manufacturing a Customized Handle of every young child or people with special needs to improve oral health for those patients by relying on themselves with an effectively way.

DETAILED DESCRIPTION:
Participants will be examined to ensure that the participants have met the sample entry criteria, then the participants will be randomly assigned to four groups each one according to a group:

1. A group of healthy children using conventional toothbrush (12 children).
2. A group of healthy children using toothbrush with Customized Handle (12 children).
3. A group of children with Down syndrome using conventional toothbrush (12 children).
4. A group of children with Down syndrome using toothbrush with Customized Handle (12 children).

Secondly,

1. Researcher will take an impression of the child hand grasp silicon impression material.
2. Researcher will scan the impression with a model scanner and copy it to the computer, then convert it -through a specialized program- to a 3D analog.
3. The program will print the digital analog via the 3D printer using Poly Lactic Acid compound and convert it into a model similar to the patient hand grasp, this model has a place to put the toothbrush.

Third, Brushing instructions:

1. The researcher will teach the participants how to brush by using (tell-show -do) technique.
2. The brushing method that will be used is the modified Stillman technique.
3. Brushing duration must be at least 3 minutes.
4. The brushing must be twice a day.
5. The amount of toothpaste is pea size.

Finally, Mechanism of examination and follow up:

After apply the plaque disclosing solution on the teeth with a bond brush, the plaque will be evaluated with Turesky Modification Quigley-Hein Plaque Index, checking on the buccal and lingual surfaces of all the teeth existing in the participant's mouth.

The participants will be observed in the same day, before and after brushing, and after one week and three weeks

ELIGIBILITY:
Inclusion criteria:

* Ages between 6-9 years old.
* Participant must have at least 10 teeth free from dental caries on both buccal and lingual surfaces of the teeth.
* TMQHPI is at least 2.
* Cooperative participant (Positive according to Frankel's behavioral rating scale).
* Parents' consent.
* Participant with down syndrome must have been diagnosed by specialist.

Exclusion criteria:

* Children undergoing orthodontic treatment.
* Allergic to any of the toothpaste ingredient used the study.
* Participant used any toothbrush other than the conventional brush before.
* Healthy children Participant with systemic diseases
* Excluding children with Down syndrome who suffer from chronic weakness such as epilepsy or taking medications continuously.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Line B Droubi, DDs, Principal Investigator — MSc student in Pedodontics, University of Damascus; Mohannad G Laflouf, Phd, Study Director — Professor of Pedodontics, Department of Pedodontics, University of Damascus
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reeson MG, Jepson NJ. Customizing the size of toothbrush handles for patients with restricted hand and finger movement. J Prosthet Dent. 2002 Jun;87(6):700. doi: 10.1067/mpr.2002.120840. No abstract available. PMID 12131899
- [Background] Kammers AC, Zanetti AL, Lacerda TE, Aroca JP, Camilotti V, Mendonca MJ. Toothbrush Handles Individually Adapted for Use by Elderly Patients to Reduce Biofilm on Complete Dentures: A Pilot Study. J Clin Diagn Res. 2015 May;9(5):ZC94-7. doi: 10.7860/JCDR/2015/11261.5975. Epub 2015 May 1. PMID 26155573

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Children Using Toothbrush With Customized Handle | Healthy Children Using Conventional Toothbrush | Children With Down Syndrome Using Conventional Toothbrush | Children With Down Syndrome Using Toothbrush With Customized Handle
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Children Using Conventional Toothbrush | Healthy Children Using Toothbrush With Customized Handle | Children With Down Syndrome Using Conventional Toothbrush | Children With Down Syndrome Using Toothbrush With Customized Handle | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 7 (.9) | 7 (.7) | 7.7 (.9) | 7.4 (1.1) | 7.2 (.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 7 | 26
  Male | 6 | 5 | 6 | 5 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 12 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Clinical Plaque Evaluation of Healthy Children and Down Syndrome of Both Groups at the Baseline
Description: Plaque scores will be assessed with Turesky Modification of the Quigley-Hein Plaque Index (TMQHPI). Plaque will be detected using plaque disclosing agent. In this index the plaque is evaluated and revealed on the buccal and lingual non-restored surfaces of the teeth on a scale of 0 to 5. Where 0 means no plaque presence which is considered as a perfect state, 1 separated ﬂecks of plaque at the cervical margin, 2 a thin continuous back of plaque (up to 1 mm) at the cervical margin, 3 a band of plaque wider than 1 mm but covering less than one-third of the side of the crown of the tooth, 4 plaque covering at least one-third but less than two-thirds of the side of crown of the tooth and finally 5 is considered as the worst state by plaque covering two-thirds or more of the side of the crown of the tooth. All teeth are assessed. The final outcome is determined by an index of the entire mouth by dividing the total score by the number of surfaces examined.
Time Frame: Baseline: Pre-brushing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Children Using Toothbrush With Customized Handle | Healthy Children Using Conventional Toothbrush | Children With Down Syndrome Using Conventional Toothbrush | Children With Down Syndrome Using Toothbrush With Customized Handle
Number analyzed (Participants) | 12 | 12 | 12 | 12
score on a scale | 3.05 (.48) | 3.19 (.5) | 3.63 (.29) | 3.41 (.25)

2. Primary Outcome: Clinical Plaque Evaluation of Healthy Children and Down Syndrome of Both Groups After Brushing
Description: as for outcome 1
Time Frame: Post-brushing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Children Using Conventional Toothbrush | Healthy Children Using Toothbrush With Customized Handle | Children With Down Syndrome Using Conventional Toothbrush | Children With Down Syndrome Using Toothbrush With Customized Handle
Number analyzed (Participants) | 12 | 12 | 12 | 12
score on a scale | 1.7 (.68) | .96 (.29) | 2.69 (.45) | .97 (.35)

3. Secondary Outcome: Clinical Plaque Evaluation of Healthy Children and Down Syndrome of Both Groups After a Week
Description: as for outcome 1
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Children Using Conventional Toothbrush | Healthy Children Using Toothbrush With Customized Handle | Children With Down Syndrome Using Conventional Toothbrush | Children With Down Syndrome Using Toothbrush With Customized Handle
Number analyzed (Participants) | 12 | 12 | 12 | 12
score on a scale | 1.41 (.39) | .38 (.43) | 2.23 (.54) | .52 (.21)

4. Post Hoc Outcome: Clinical Plaque Evaluation of Healthy Children and Down Syndrome of Both Groups After Three Weeks
Description: as for outcome 1
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Children Using Toothbrush With Customized Handle | Healthy Children Using Conventional Toothbrush | Children With Down Syndrome Using Conventional Toothbrush | Children With Down Syndrome Using Toothbrush With Customized Handle
Number analyzed (Participants) | 12 | 12 | 12 | 12
score on a scale | .14 (.27) | 1.21 (.47) | 1.91 (.58) | .26 (.1)

ADVERSE EVENTS:
Time Frame: Throw study completion.Plaque accumulation was evaluated at four times 1- Pre-brushing at baseline. 2- Post-brushing at baseline. 3- 1 week from baseline 4- 3 weeks from baseline .
Description: Serious or other non-serious adverse events were not collected in the current trial.
Arm/Group | Healthy Children Using Toothbrush With Customized Handle | Healthy Children Using Conventional Toothbrush | Children With Down Syndrome Using Conventional Toothbrush | Children With Down Syndrome Using Toothbrush With Customized Handle
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Base line between normal children group and down children group can not be achieved easily, yet it can be compared later after a week and three weeks and give some valuable information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT04845633/Prot_SAP_000.pdf